CLINICAL TRIAL: NCT06786780
Title: A Single-Arm, Single-Center, Phase II Study to Evaluate the Predictive Value of Organoids for Radiotherapy and Chemotherapy Efficacy in Cervical Cancer
Brief Title: Establishment and Validation of Prediction Model of Simultaneous Chemoradiotherapy for Cervical Cancer Organoids
Acronym: ECCO
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Chongqing University Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CQGOG0115; BJHA-CRP-079 (Other Grant/Funding Number: Beiing Health Alliance Charitable Foundation，China)
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-12

CONDITIONS: Cervical Cancer Treated with Pelvic Radiotherapy; Cervical Cancers
Keywords: Cervical cancer; Concurrent chemoradiotherapy; organoid
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin

STUDY DESIGN:
Intervention Model Description: By extracting tumor tissues from cervical squamous cell carcinoma, adenocarcinoma, small cell carcinoma, neuroendocrine carcinoma, clear cell carcinoma, intestinal-type adenocarcinoma, mesonephric adenocarcinoma, and mucinous adenocarcinoma, cervical cancer organoids are constructed. These organoids undergo concurrent chemoradiotherapy experiments, and the results are compared with clinical efficacy to construct a model for predicting clinical concurrent chemoradiotherapy outcomes, which is then used to validate the efficacy of clinical concurrent chemoradiotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: treatment arm (Experimental): Participants receive concurrent chemoradiotherapy, including external beam radiation therapy (EBRT) or brachytherapy. Cisplatin is administered at a dose of 100mg/m² every three weeks, with two doses given during the radiotherapy period, totaling a dose of 200mg/m², or cisplatin at a dose of 40mg/m² once a week, for approximately six weeks of treatment, totaling a dose of 240mg/m². Treatment continues until intolerable toxicity occurs or the investigator determines that the subject can no longer benefit. Before concurrent chemoradiotherapy, cervical cancer tumor tissue or ascites are collected to construct organoids for concurrent chemoradiotherapy experiments. After disease progression, cervical cancer tissue or ascites are collected to construct organoids for drug screening experiments.
  Interventions: Combination Product: Drug: Cisplatin

INTERVENTIONS:
Combination Product: Drug: Cisplatin — Organoids were constructed prior to simultaneous radiochemical therapy

SUMMARY:
This is a single-arm, single-center, open-label, Phase II study aimed at assessing the efficacy of organoids in predicting the response to radiotherapy and chemotherapy in cervical cancer

DETAILED DESCRIPTION:
By constructing cervical cancer organoids, establishing a radiochemotherapy prediction model based on organoids, and exploring radiotherapy resistance-related molecules as new therapeutic targets for locally advanced cervical cancer, the feasibility and effectiveness are assessed. Utilizing the constructed model for molecular mechanism discussions and effective drug screening, new avenues for the treatment of cervical cancer patients with radiochemotherapy resistance are sought.

ELIGIBILITY:
Inclusion Criteria:

Able to understand and voluntarily sign written informed consent.

1. Women aged ≥18 years at the time of study entry.
2. Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0-2.Life expectancy ≥12 weeks.
3. Histologically confirmed cervical cancer.
4. Histologically-confirmed squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma，villous duct carcinoma, invasive mucinous multilayer carcinoma, gastric adenocarcinoma, mesrenal duct carcinoma, clear cell carcinoma, serous carcinoma, endometrioid adenocarcinoma and small cell carcinoma，Intestinal-type adenocarcinoma of the cervix;
5. At least one measurable tumor lesion according to RECIST v1.1 criteria.
6. Available archived tumor tissue samples or recent biopsies.
7. Adequate organ function.
8. For fertile women with negative serum pregnancy and effective contraception within 7 days before administration (until 120 days after the last administration of the study drug and at least 180 days after radiotherapy)

Exclusion Criteria:

1. Subject with other active malignancies within 2 years prior enter the study.
2. Subject who cannot receive brachytherapy.
3. Active or prior documented autoimmune disease that may relapse.
4. History of interstitial lung disease or noninfectious pneumonitis.
5. Subject with the clinically significant cardio-cerebrovascular disease.
6. History of severe hypersensitivity reactions to other mAbs.
7. Prior allogeneic stem cell transplantation or organ transplantation.
8. Subjects who require systemic treatment with glucocorticoid (>10 mg/day of prednisone or equivalent glucocorticoid) or other immunosuppressive agents within 14 days prior enter the study.
9. Receipt of live attenuated vaccines within 30 days prior to the first dose of the study drug.
10. Prior exposure to any experimental antitumor vaccines, or any agent targeting T-cell costimulation or immune checkpoint pathways (eg, anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4, anti-CD137 or anti-OX40 antibody, etc).
11. Any condition that, in the opinion of the Investigator, would interfere with the evaluation of the study drug or interpretation of subject safety or study results.

    -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
ORR assessed by Investigator | Up to 1 years
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR per RECIST v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Ling Long, PhD, Principal Investigator — Chongqing University Cancer Hospital
Locations (1):
- Chongqing university Cancer Hospital, Chongqing, China, China

IPD SHARING:
Plan to Share IPD: No
Involving patient privacy